CLINICAL TRIAL: NCT05380622
Title: CHART Study of Coronary CT Angiography to Predict Imaging and Cardiovascular Outcomes in Patients With Coronary Artery Disease
Brief Title: CHART Study of Coronary CT Angiography in Coronary Artery Disease
Acronym: CHART-VISION
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHART-20220510
Record Dates: First submitted 2022-05-10; First posted 2022-05-19 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without ICA or deferral of PCI after ICA group: Patients didn't undergo invasive coronary angiography (ICA) or with a vessel determined to defer revascularization.
  Interventions: Diagnostic Test: Coronary CT angiography
- PCI group: Patients with a vessel that undergo percutaneous coronary intervention (PCI)
  Interventions: Diagnostic Test: Coronary CT angiography

INTERVENTIONS:
Diagnostic Test: Coronary CT angiography — Coronary CT angiography (CCTA) will be performed according to standard protocol and measurement of fractional flow reserve (FFR) or other physiological indices will be at the at the discretion of the physicians in charge.
  Stenosis and plaque features, disease patterns, hemodynamic parameters, and fat metrics on CCTA will be analyzed blindly in the core lab.

SUMMARY:
In a cohort of patients referred to coronary computed tomography angiography (CCTA), the investigators aim:

1. To describe the natural history of the coronary atherosclerotic plaque development and progression or regression, as well as the plaque characterization and phenotypes over time by CCTA among deferred coronary lesions
2. To explore the precursors of plaques leading to acute coronary syndrome (ACS) or chronic coronary syndrome (CCS) in deferred coronary lesions
3. To investigate prognostic implication of qualitative and quantitative plaque analysis of stenosis and plaque features, disease patterns, hemodynamic parameters, and fat metrics on CCTA along with physiologic assessment
4. To investigate the effects of different treatment strategies according to stenosis and plaque features, fat metrics on CCTA along with physiologic assessments.

DETAILED DESCRIPTION:
Invasive physiologic indices such as fractional flow reserve (FFR) are used to define ischemia-causing stenosis and guide percutaneous coronary intervention (PCI) in the clinical practice. FFR-guided PCI has been proven to improve clinical outcomes, however, a substantial proportion of patients continue to experience clinical events. The ISCHEMIA trial showed that invasive therapy did not improve prognosis in patients with moderate to severe ischemia compared to optimal medical therapy. Besides, a recent study implied that even in vessels with FFR>0.80, those have lesions with high-risk plaque characteristics (HRPC) demonstrated worse clinical outcomes. This might be not unexpected since previous evidence from postmortem studies demonstrated that unstable atherosclerotic plaques are prone to rupture and trigger adverse cardiovascular events.

In recent years, advances in imaging analysis made it possible to conduct novel measurements such as pericoronary inflammation or epicardial fat metrics and lesion-specific or vessel-specific hemodynamic parameters derived from CCTA (such as fractional flow reserve by CCTA [CT-FFR]) as well as the coronary disease patterns defined by physiologic distribution (predominant focal versus diffuse disease defined by CCTA derived pullback pressure gradient index) and local severity (presence versus absence of major gradient defined by CCTA-derived FFR gradient per unit length [dCT-FFR/ds]) of coronary atherosclerosis.

However, the relationship of these parameters and the combination of these indices on clinical outcomes has not been fully understood. Furthermore, though it has been known that high-risk plaques are related with worse outcomes even no significant blood flow impairment induced, best treatment strategy for these lesions remains unclear.

In this regard, the aims of this study are multiple, all the treatment strategies are at the discretion of the physicians in charge. For patients without further invasive angiography performed after CCTA or deferred for revascularization after invasive angiography with/without physiology or imaging assessments, the investigators will investigate coronary atherosclerotic plaque development and progression or regression, as well as the plaque characterization and phenotypes over time by CCTA, and to explore the precursors of plaques leading to acute coronary syndrome (ACS) or chronic coronary syndrome (CCS); for those with received revascularization, the investigators will investigate the prognostic value of CCTA based comprehensive analysis of coronary in combination with physiologic assessment. In all patients, the effects of different treatment strategies according to stenosis and plaque features, fat metrics as well as physiologic assessments will be investigated.

CHART is a study group called Chinese Non-invasive Cardiovascular Imaging and Physiology Study Group, the current study will be conducted by CHART and by invitation in multiple Chinese centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for CCTA.
* Qualified patients who have signed a written informed consent form.

Exclusion Criteria:

* Left ventricular ejection fraction < 35%
* Acute ST-elevation myocardial infarction within 72 hours or previous coronary artery bypass graft surgery
* Abnormal epicardial coronary flow (TIMI flow < 3)
* Planned coronary artery bypass graft surgery after diagnostic angiography
* Poor quality of CCTA or other reasons by core lab that are unsuitable for plaque, physiological or fat analysis
* Patients with a stent in the target vessel

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for CCTA.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of high-risk plaques | 30 days
  Frequency (%) of occurrence of high-risk plaque morphologic features (Housfield Unit[HU]<30, Remodelling Index > 1.1, napkin-ring sign, spotty calcium, minimal lumen area[MLA]<4mm2 & plaque burden[PB]≥70%), physiologic diffuse disease, inflammation by high fat attenuation index (FAI)
Change in total plaque volume (adjusted by vessel volume) and plaque composition detected by follow up CCTA | up to 5 years after index procedure
  Change in total plaque volume (adjusted by vessel volume) and plaque composition detected by follow up CCTA
Change in WSS detected by follow up CCTA | up to 5 years after index procedure
  Change in hemodynamic parameter of wall shear stress (WSS) detected by follow up CCTA
Change in APS detected by follow up CCTA | up to 5 years after index procedure
  Change in hemodynamic parameter of axial plaque stress (APS) detected by follow up CCTA
Change in SSI detected by follow up CCTA | up to 5 years after index procedure
  Change in stenosis susceptibility index (SSI) detected by follow up CCTA
Change in hemodynamic parameters delta fractional flow reserve detected by follow up CCTA | up to 5 years after index procedure
  Change in hemodynamic parameters delta fractional flow reserve detected by follow up CCTA
Change in physiological pattern by PPG derived by follow up CCTA | up to 5 years after index procedure
  Change in physiological pattern by pullback pressure gradient (PPG) derived by follow up CCTA
Change in dCT-FFR/ds detected by follow up CCTA | up to 5 years after index procedure
  Change in dCT-FFR/ds detected by follow up CCTA
Change in CT-FFR | up to 5 years after index procedure
  Change in fractional flow reserve by CCTA
Change in peri-coronary adipose tissue assessed by follow up CCTA | up to 5 years after index procedure
  Change in peri-coronary adipose tissue assessed by follow up CCTA
CCTA-derived features associated with precursors of ACS or CCS | up to 5 years after index procedure
  CCTA-derived features associated with precursors of ACS or CCS
Adverse cardiovascular event according to stenosis and plaque features, disease patterns, hemodynamic parameters, and fat metrics on CCTA along with physiologic assessment | up to 5 years after index procedure
  A composite of cardiac death, vessel-related myocardial infarction (MI), or vessel-related ischemia-driven revascularization.
Adverse cardiovascular event according to different treatment strategies according to stenosis and plaque features, fat metrics on CCTA along with physiologic assessments. | up to 5 years after index procedure
  A composite of cardiac death, vessel-related myocardial infarction (MI), or vessel-related ischemia-driven revascularization.

SECONDARY OUTCOMES:
Anginal status | up to 5 years after index procedure
  Change in Health Related Quality of Life (HRQL)
Number of anti-anginal medication prescribed | up to 5 years after index procedure
  Number of anti-anginal medication prescribed
Clinical predictors of events | up to 5 years after index procedure
  To find out the models with baseline characteristics including age, sex, cardiovascular risk factors and so on with the highest area under curve to predict a composite of cardiac death, vessel-related myocardial infarction (MI), or vessel-related ischemia-driven revascularization.
Prognostic value of CCTA defined anatomy and plaque characterization | up to 5 years after index procedure
  Prognostic value of CCTA defined anatomy including diameter stenosis, area stenosis and plaque characterization including plaque components, physiological on blood flow, diffuseness and inflammation.
Prognostic value of WSS | up to 5 years after index procedure
  Prognostic value of WSS
Prognostic value of APS | up to 5 years after index procedure
  Prognostic value of APS
Prognostic value of SSI | up to 5 years after index procedure
  Prognostic value of SSI
Prognostic value of delta CT-FFR | up to 5 years after index procedure
  Prognostic value of delta CT-FFR
Prognostic value of pull pressure gradient | up to 5 years after index procedure
  Prognostic value of pull pressure gradient
Prognostic value of dCT-FFR/ds | up to 5 years after index procedure
  Prognostic value of dCT-FFR/ds
Prognostic value of per-coronary adipose tissue | up to 5 years after index procedure
  Prognostic value of per-coronary adipose tissue derived fat attenuation index and other radiomics features.
Prognostic value of integrated CCTA based lesion anatomy, plaque characterization, hemodynamic parameters, physiological patterns and per-coronary adipose tissue for ACS | up to 5 years after index procedure
  Comparison of outcome discrimination ability.
Prognostic value of integrated CCTA based lesion anatomy, plaque characterization, hemodynamic parameters, physiological patterns and per-coronary adipose tissue for cardiovascular events | up to 5 years after index procedure
  Comparison of outcome discrimination ability.
Relationship among CT-derived plaque qualification and quantification, and CT-defined pericoronary and epicardial fat metrics with physiological assessments. | up to 5 years after index procedure
  Association among CCTA parameters (including diameter stenosis, area stenosis, plaque components) and physiologic indices (CT-FFR, PPG, delta-FFR, dCT-FFR/ds).

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Study Chair — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided